CLINICAL TRIAL: NCT00999687
Title: Evaluation of the Efficacy and Safety of Indigo Naturalis Oil Extract on Psoriatic Nails
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yin-ku Lin, Chief of department of traditional Chinese medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG280191
Record Dates: First submitted 2009-10-20; First posted 2009-10-22 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Nail Psoriasis
Keywords: Nail psoriasis; Indigo naturalis
MeSH Terms: interventions — Oils; Olive Oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indigo naturalis extract in oil (Experimental): Indigo naturalis extract in oil (INEO) was applied to the fingernails of one bilateral hand (experimental group) twice daily for the first 12 weeks. INEO was applied to all affected nails on both hands twice daily for another 12 weeks.
  Interventions: Drug: Indigo Naturalis Extract in Oil
- Olive oil (Placebo Comparator): Olive oil was applied to the fingernails of the contra-lateral hand (control group) twice daily for the first 12 weeks. INEO was applied to all affected nails on both hands twice daily for another 12 weeks.
  Interventions: Drug: Indigo Naturalis Extract in Oil; Other: Olive Oil

INTERVENTIONS:
Drug: Indigo Naturalis Extract in Oil — Indigo naturalis extract in oil (INEO) was applied to the fingernails of one bilateral hand (experimental group) twice daily for the first 12 weeks. INEO was applied to all affected nails on both hands twice daily for another 12 weeks
  Other Names: INEO
Other: Olive Oil — Olive oil was applied to the fingernails of the contra-lateral hand (control group) twice daily for the first 12 weeks. INEO was applied to all affected nails on both hands twice daily for another 12 weeks.
  Arms: Olive oil

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of indigo naturalis oil extract in treating nail psoriasis.

DETAILED DESCRIPTION:
Nail psoriasis treatment is notoriously difficult. While indigo naturalis has been demonstrated safe and effective in treating skin psoriasis, its effect on nail psoriasis remains unverified.

ELIGIBILITY:
Inclusion criteria:

1. adults aged between 20 and 65 years
2. received a diagnosis of nail psoriasis with at least one year history based on clinical assessment by two dermatologists and failure of topical systemic Chinese herbal anti-psoriasis therapy for fingernail psoriasis.
3. Female patients of childbearing age agreed to continue using birth control measures for the duration of the study.

Exclusion criteria:

1. Patients had non-plaque (i.e., pustular, guttate, or erythrodermic) or drug-induced forms of psoriasis, total body surface involvement of more than 60%
2. a history of allergy to indigo naturalis, or with onychomycosis or any fingernail infection.
3. Patients have received systemic therapy within four weeks before enrollment
4. Patients have received phototherapy within three weeks, or topical psoriasis agents within two weeks.
5. Using medications which affect psoriasis during the study and unwillingness to comply with study protocol.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Ku Lin, MD. PhD., Principal Investigator — Chang Gung Memorial Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from ambulatory department of Chang Gung Memorial Hospital, in northern Taiwan between November 2009 and May 2011.
Pre-assignment Details: 35 participants recruited and screened, 4 excluded (3 did not meet the eligibility criteria and 1 refused participation).
Groups:
- All Participants (Indigo Naturalis Oil Extract /Olive Oil): In all participants, indigo naturalis oil extract (INOE) was applied to the fingernails of one bilateral hand (experimental group) and olive oil was applied to the fingernails of the contralateral hand (control group) twice daily for 12 weeks. The randomization process was conducted by block randomization method with 1:1 ratio. After 12 weeks, olive oil treatment was discontinued and INOE was applied to both hands twice daily for another 12 weeks.
Period: First Intervention
Arm/Group | All Participants (Indigo Naturalis Oil Extract /Olive Oil)
Started | 31 (16 used the INOE on the right hand,15 used the INOE on the left hand.)
Completed | 30
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Second Intervention
Arm/Group | All Participants (Indigo Naturalis Oil Extract /Olive Oil)
Started | 30 (From week 13 to 24, all participants applied INOE to both hands twice daily.)
Completed | 27
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants (Indigo Naturalis Oil Extract /Olive Oil): In all participants, indigo naturalis oil extract was applied to the fingernails of one bilateral hand (experimental group) and olive oil was applied to the fingernails of the contralateral hand (control group) twice daily for 12 weeks. The randomization process was conducted by block randomization method with 1:1 ratio. After 12 weeks, olive oil treatment was discontinued and indigo naturalis oil extract was applied to both hands twice daily for another 12 weeks.
Arm/Group | All Participants (Indigo Naturalis Oil Extract /Olive Oil)
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Single-Hand Nail Psoriasis Severity Index (NAPSI)and in the Modified Target NAPSI for the Single Most Severely Affected Nail of Each Hand at Week 12.
Description: The nail is divided by imaginary horizontal and longitudinal lines into quadrants. Each nail is given a score for nail bed psoriasis (0-4) and nail matrix psoriasis (0-4) depending on the presence of any of the features of nail psoriasis in that quadrant. The NAPSI score evaluates presence of signs in the nail bed (of onycholysis, splinter hemorrhages, nail bed discoloration, and subungual hyperkeratosis) and on the nail matrix (pitting, leukonychia, red spots in the lunula and nail plate crumbling) in all 10 fingernails, providing a minimal score of 0 and a maximum of 80. This study is an intra-patient side-to-side comparison, it measures nail disease on a single hand. All 5 fingers in each group were scored providing a maximum score of 40 and a minimal of 0. The modified target NAPSI score for the target nail scores severity of nail matrix and nail-bed psoriasis from 0 (no sign) to 3 (severe involvement) in each nail quadrant, providing a maximum score of 96 and a minimal of 0.
Time Frame: Baseline and Week 12
Population: Higher values represent a worse outcome. For example, a higher score at baseline and a lower score after treatment represent an improvement.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Experimental Group: Using Indigo Naturalis Oil Extract (INOE) from week 0 to week 24.
- Control Group: Using Olive Oil from week 0 to week 12, then change to Indigo Naturalis Oil Extract (INOE) from week 13 to week 24.
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 30 | 30
units on a scale
  Change from Baseline in Single-Hand NAPSI | -10.9 (6.0) [-13.30 to -8.52] | -4.9 [-6.95 to -2.78]
  Change from Baseline in Modified-Target NAPSI | -8.1 [-9.97 to -6.23] | -2.2 [-3.76 to -0.57]

2. Primary Outcome: Change From Baseline in Single-Hand Nail Psoriasis Severity Index (NAPSI)and in the Modified Target NAPSI for the Single Most Severely Affected Nail of Each Hand at Week 24.
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Control Group: Using Olive Oil from week 0 to week 12, then transfer to Indigo Naturalis Oil Extract from week 13 to week 24
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 27 | 27
units on a scale
  Change from Baseline in Single-Hand NAPSI | -13.4 [-16.40 to -10.50] | -11.6 [-14.20 to -9.05]
  Change from Baseline in Modified-Target NAPSI | -10.6 [-12.60 to -8.54] | -8.0 [-9.74 to -6.34]

ADVERSE EVENTS:
Time Frame: Baseline and Week 24
Groups:
- All Participants (Indigo Naturalis Oil Extreact/Olive Oil): Experimental group: randomized to receive Indigo Naturalis Oil Extract first; Control group: randomized to receive Olive Oil first.
  In all participants, indigo naturalis oil extract was applied to the fingernails of one bilateral hand (experimental group) and olive oil was applied to the fingernails of the contralateral hand (control group) twice daily for 12 weeks. The randomization process was conducted by block randomization method with 1:1 ratio. After 12 weeks, olive oil treatment was discontinued and indigo naturalis oil extract was applied to both hands twice daily for another 12 weeks.
Arm/Group | All Participants (Indigo Naturalis Oil Extreact/Olive Oil)
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes